CLINICAL TRIAL: NCT04237103
Title: Efficacy and Tolerance of the Combination of Methotrexate and Phototherapy Versus Phototherapy in Adults With Progressive Vitiligo: a Randomized Double-blind Prospective Study
Brief Title: Combination of Methotrexate and Phototherapy Versus Phototherapy in Adults With Progressive Vitiligo
Acronym: METVI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUBX 2017/44
Record Dates: First submitted 2019-05-23; First posted 2020-01-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Vitiligo
Keywords: vitiligo; pigmentation; phototherapy; methotrexate
MeSH Terms: conditions — Vitiligo | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: Methotrexate taken orraly once a weekcombination with UVB TL01 in a population of adult patients with progressive vitiligo
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study was performed double blind. MTX will be repackaged in capsules and will look the same as placebo capsules. These capsules are packaged in vials whose labeling allows the maintenance of the blind.
  The flasks are numbered in a corresponding list established by biostatistician study which specifies processing to be put in each bottle according to the number.
  At each visit (inclusion and monitoring), the patient will be assigned as many lots of numbers needed to reach the next visit (2 or 4).
  Only Methods Center (USMR) and Pharmacy of Bordeaux University Hospital have the correspondence between the number of treatment and nature. At no time during the study, the investigator (s) and patients will not have access to this list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methotrexate (Experimental): Methotrexate once a week orally for 8 months in conjunction with narrow band UVB phototherapy starting 2 months after Methotrexate therapy for 6 months.
  Interventions: Drug: Methotrexate
- placebo (Placebo Comparator): Placebo once a week orally for 8 months in conjunction with narrow band UVB phototherapy starting 2 months afterplacebo therapy, for 6 months.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Methotrexate — oral capsules taken once a week
  Other Names: narrow-band UVB phototherapy
  Arms: methotrexate
Drug: Placebos — Administered identically to the experimental group
  Other Names: narrow-band UVB phototherapy
  Arms: placebo

SUMMARY:
This is a phase 2, randomized, double blind, multicenter study evaluating the efficacy and safety of the combination of methotrexate plus UVB TL01 in vitiligo.

DETAILED DESCRIPTION:
Treatment Strategy: Multicentric, parallel double blind randomized phase 2 prospective study comparing MTX taken orally once a week + narrowband UVB TL01 versus placebo + narrowband UVB TL01 Follow-up of the study: patients included in this study will start MTX 2 months before starting narrowband UVB TL01. Phototherapy will be performed twice a week during 6 months. Follow-up visit will be done at month 2, 4 and month 8. Phone calls to the patient will be done at month 6

ELIGIBILITY:
Inclusion Criteria:

* Subject male or female age over 18 years old
* Diagnosis of non-segmental (symmetrical) vitiligo with body surface area ≥10%
* Active non-segmental vitiligo defined by Non-segmental vitiligo with new patches or extension of old lesions during the last 6 months AND Presence of hypochromic aspect under Wood's lamp examination and/or perifollicular hypopigmentation under Wood's lamp examination.
* Signed informed consent document
* Male patients agreeing to use a reliable method of birth control during the study i. e. preservative and for at least 6 months following the last dose of investigational product, the patient's partner treated by methotrexate must be notified of the teratogenic risk of methotrexate and should be under effective contraception throughout the study and for at least 6 months following the last dose of investigational product.
* Women of childbearing potential who are negatively tested for pregnancy and agree to use a reliable method of birth control (every month) or remain abstinent during the study and for at least 6 months following the last dose of investigational product. Methods of contraception considered acceptable include oral contraceptives, contraceptive patch, intrauterine device, vaginal ring
* Patient registered to the French Social Security

Exclusion Criteria:

* Segmental or mixed vitiligo
* Patients who have known active liver disease (with the exception of a simple liver steatosis, transaminases and/or alkaline phosphatases > 2 ULM ) or history of liver disease in the past 2 years, whatever the related diagnosis but which could interfere with MTX safety and according to the summary of the SmPC.
* Intake of restricted medications (cf section VIII.5.) or other drugs considered likely to interfere with the safe conduct of the study, as assessed by the investigator and according to the Summary of the Product Characteristics (SmPC), including any drug intakes that could interfere with methotrexate metabolism or that could enhance liver and /or hematologic toxicity and according to the SmPC
* Patient with evidence or positive test for HIV, Hepatitis C virus, Hepatitis B virus (patients who are negative for hepatitis B surface antigen but positive for anti-hepatitis B anti body (HBsAb+ and HBcAb+) and negative for serum HBV DNA may participate in the study
* High alcohol intake defined as more than 60 g of daily intake (approx daily intake of 0.5 l of wine or equivalent),
* Patients who have a known allergy or hypersensitivity to MTX
* Patients who have a known serious adverse event to MTX prior to the trial leading to MTX discontinuation in the past
* Presence of significant hematologic or renal disorder or abnormal laboratory values at screening that, in the opinion of the investigator is associated with an unacceptable risk to the patient to participate in the study
* Clinical laboratory test results at screening that are outside a normal reference rating for the population and are considered clinically significant, or/and have any of the following specific abnormalities:
* Total white blood cell count <3G/L
* Neutrophil count < 1.5 G/l
* Lymphocytes count < 0.5G/l
* Platelet count < 100 G/l
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>3 times the upper limit of normal (ULM)
* Hemoglobin <8.5g/dL (85.0 g/L)
* Creatinine clearance <40ml/min (Cockcroft formula)
* For women: pregnant or breast feeding
* Patients who have an active or serious infection or history of infections (bacterial, viral, fungal or mycobacteria), requiring hospitalization or intra venous anti-infectives infusion within 4 weeks prior to the baseline,
* Patients who have primary or secondary active immunodeficiency
* Patients who had live vaccine administration within 4 weeks prior to baseline
* Patients who had already been treated by at least 250 sessions of phototherapy - Patients who have any current or active cancer (with the exception of patient with successfully treated with in situ cervix carcinoma)
* Patients who had history of malignancy within 5 years prior to the trial that could contraindicate the use of an immunosuppressant
* Patients who will not be available for protocol which require study visits or procedures
* Patients who is not affiliated to the French Social Security system
* Patients unable to give informed consent and/or comply with all required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Score with VASI formule | month 8
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.

SECONDARY OUTCOMES:
Score with VASI formule | month 4
  Change in percentage of repigmented Surface area 4 months after-inclusion, by using the VASI score at M4.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
Number of Adverse Events (AE) and serious adverse events (SAE), as well as the proportion of discontinuation due to AEs and/or SAEs | Month 8
  AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related, that occurs after a subject provides informed consent. Abnormal laboratory values or test results occurring after informed consent constitute AEs only if they induce clinical signs or symptoms, are considered clinically meaningful, require therapy, or require changes in the study drug.
Evaluation of score Vitiligo European Task Force (VETF) | Month 4
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score Vitiligo European Task Force (VETF) | Month 8
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score of the Vitiligo Extent Score (VES) | Month 4
  Variation in percentage of the Vitiligo Extent Score (VES). The VES score is used to assess the severity and extent of vitiligo. Using the VES calculator www.vitiligo-calculator.com, investigator choose the pictures that best represent the patient's skin lesions and then the percentage of depigmented area is calculated.
Evaluation of score of the Vitiligo Extent Score (VES) | Month 8
  Variation in percentage of the Vitiligo Extent Score (VES). The VES score is used to assess the severity and extent of vitiligo. Using the VES calculator www.vitiligo-calculator.com, investigator choose the pictures that best represent the patient's skin lesions and then the percentage of depigmented area is calculated.
Evaluation of score of the Dermatology Life Quality Index (DLQI) | Month 4
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) | Month 8
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 3.
Evaluation of the score of the Skindex 29 | Month 4
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Skindex 29 | Month 8
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Vitiligo Impact Scale (VIP) | Month 4
  Variation of the score of the Vitiligo Impact Scale (VIP). Vitiligo Impact Scale is a 2-item instrument, each item scored from 0 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 145
Evaluation of the score of the Vitiligo Impact Scale (VIP) | Month 8
  Variation of the score of the Vitiligo Impact Scale (VIP). Vitiligo Impact Scale is a 2-item instrument, each item scored from 0 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 145
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | Day 1
  Epression of MxA CD3, CD4, CD8, CXCR3, CCR6, CXCL9, 10, 11, CCL20 et HSP70
Evaluation of skin inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | Day 1
  Expression of IFN-α, TNF-α, IFN-γ, IL-17, IL-22, CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, HSP70 soluble

CONTACTS AND LOCATIONS:
Overall Officials: Julien SENESCHAL, MD, PhD, Principal Investigator — University of Bordeaux
Locations (4):
- France (4):
  - Service de Dermatologie - Hôpital Saint-André, Bordeaux, Bordeaux
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier de Périgueux, Périgueux
  - Service de Dermatologie - CHU de Toulouse - Hopital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF